CLINICAL TRIAL: NCT03212222
Title: How Does Visual Acuity Assessment Using the Peek Acuity Application Compare to the Standard Exam in the Clinic?
Brief Title: Cell Phone Application for Vision Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Pro00083577
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2018-09

CONDITIONS: Visual Impairment
Keywords: screening; cell phone application
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: Patient randomly assigned to either be screened first with standard clinic technique or cell phone application. Patient is then screened with other method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peek Acuity Screening (Experimental): Cell phone application to be used for visual acuity screening.
  Interventions: Other: Peek Acuity
- Standard Visual Screening (Active Comparator): Standard visual acuity screening administered at Duke University Eye Center regarded as the gold standard.
  Interventions: Other: Standard Visual Screening

INTERVENTIONS:
Other: Peek Acuity — Cell phone application for visual acuity screening
  Arms: Peek Acuity Screening
Other: Standard Visual Screening — Visual screening exam conducted in Duke University Eye Center
  Arms: Standard Visual Screening

SUMMARY:
The purpose of this study is to evaluate how visual acuity assessed with Peek Acuity (a cell phone application to check visual acuity) among preschool and school-aged children 3 to less than18 years of age (1) compares to the standard visual acuity exam in the ophthalmology clinic and (2) performs as a screening test for ocular abnormalities that warrant referral for an eye exam.

DETAILED DESCRIPTION:
Current recommendations suggest that children begin visual acuity screening as early as possible with most children capable at 3 years old though some may not be able to cooperate until 4 years of age. While visual acuity screening is standard in schools and pediatric clinics, the specificity of the exams has been questioned. A number of community screening exams rely on outdated and flawed methods that may not accurately access the vision of all children. Because many children who fail these vision screenings are referred to ophthalmology clinics without a true visual acuity deficit, a more accurate but accessible, cost effective, and feasible vision screening exam is necessary. One solution is a smart phone application designed to assess visual acuity, called Peek Acuity. The application is available for android operating system and can be downloaded as a free beta from the Google Play Store. A short tutorial walks users through the application. The application displays a single letter "E" in 4 positions, 0, 90, 180, and 270 degrees (rolling "E") that does not require English comprehension. Patients are instructed to point in the direction of the arms of the "E." The examiner records the responses by swiping the screen in the direction the patient points. The application uses responses to calculate visual acuity and typical exams can be completed within 2 minutes.

In one study, Peek Acuity visual assessments have been shown to be comparable to that determined by the ophthalmology clinic in patients aged 55 years and older. This study also found that the Peek Acuity is efficient, with an average exam time of 77 seconds compared to 82 seconds using the standard Snellen eye chart.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide consent
* 3 to less than 18 years of age

Exclusion Criteria:

* Unable or unwilling to give consent
* Over 18 years of age
* Less than 3 years of age

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of screening with standard exam vs. Peek Acuity for referral to further medical management | Visit 1 (up to 30 minutes)
  Children screened positive for visual deficit by standard exam will be deemed true positives; any true positives not identified by the Peek Acuity application will be deemed false negatives. Sensitivity is calculated by true positive population divided by the sum of true positives and false negatives
Specificity of screening with standard exam vs. Peek Acuity for referral to further medical management | Visit 1 (up to 30 minutes)
  Children screened negative for visual deficit by standard exam will be deemed true negatives; any true negatives not identified by the Peek Acuity application will be deemed false positives. Specificity is calculated by true negative population divided by the sum of true negatives and false positives
Accuracy of screening with standard exam vs. Peek Acuity for referral to further medical management | Visit 1(up to 30 minutes)
  Visual acuity score determined by Peek Acuity will be compared to the score from standard exam to determine accuracy where the score from standard exam is the accepted value

SECONDARY OUTCOMES:
Efficiency of screening with standard exam and Peek Acuity | Visit 1(up to 30 minutes)
  Compare average exam time between standard exam and Peek Acuity

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Jones, Study Director — Duke University
Locations (1):
- Duke UMC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barry JC, Konig HH. Test characteristics of orthoptic screening examination in 3 year old kindergarten children. Br J Ophthalmol. 2003 Jul;87(7):909-16. doi: 10.1136/bjo.87.7.909. PMID 12812897
- [Background] Miller JM, Dobson V, Harvey EM, Sherrill DL. Cost-efficient vision screening for astigmatism in native american preschool children. Invest Ophthalmol Vis Sci. 2003 Sep;44(9):3756-63. doi: 10.1167/iovs.02-0970. PMID 12939288
- [Background] Anstice N, Spink J, Abdul-Rahman A. Review of preschool vision screening referrals in South Auckland, New Zealand. Clin Exp Optom. 2012 Jul;95(4):442-8. doi: 10.1111/j.1444-0938.2012.00713.x. Epub 2012 Apr 17. PMID 22507224
- [Background] Simons K. Preschool vision screening: rationale, methodology and outcome. Surv Ophthalmol. 1996 Jul-Aug;41(1):3-30. doi: 10.1016/s0039-6257(97)81990-x. PMID 8827927
- [Background] Schmucker C, Grosselfinger R, Riemsma R, Antes G, Lange S, Lagreze W, Kleijnen J. Diagnostic accuracy of vision screening tests for the detection of amblyopia and its risk factors: a systematic review. Graefes Arch Clin Exp Ophthalmol. 2009 Nov;247(11):1441-54. doi: 10.1007/s00417-009-1150-2. Epub 2009 Aug 11. PMID 19669781
- [Background] Alexander P, Rahi JS, Hingorani M. Provision and cost of children's and young people's eye services in the UK: findings from a single primary care trust. Br J Ophthalmol. 2009 May;93(5):645-9. doi: 10.1136/bjo.2008.149203. Epub 2008 Dec 19. PMID 19098035
- [Background] Joish VN, Malone DC, Miller JM. A cost-benefit analysis of vision screening methods for preschoolers and school-age children. J AAPOS. 2003 Aug;7(4):283-90. doi: 10.1016/s1091-8531(03)00116-2. PMID 12917617
- [Background] Bastawrous A, Rono HK, Livingstone IA, Weiss HA, Jordan S, Kuper H, Burton MJ. Development and Validation of a Smartphone-Based Visual Acuity Test (Peek Acuity) for Clinical Practice and Community-Based Fieldwork. JAMA Ophthalmol. 2015 Aug;133(8):930-7. doi: 10.1001/jamaophthalmol.2015.1468. PMID 26022921
- [Background] Committee on Practice and Ambulatory Medicine Section on Ophthalmology; American Association of Certified Orthoptists; American Association for Pediatric Ophthalmology and Strabismus; American Academy of Ophthalmology. Eye examination in infants, children, and young adults by pediatricians: organizational principles to guide and define the child health care system and/or improve the health of all children. Ophthalmology. 2003 Apr;110(4):860-5. doi: 10.1016/S0161-6420(03)00414-7. PMID 12689914
- [Derived] Zhao L, Stinnett SS, Prakalapakorn SG. Visual Acuity Assessment and Vision Screening Using a Novel Smartphone Application. J Pediatr. 2019 Oct;213:203-210.e1. doi: 10.1016/j.jpeds.2019.06.021. Epub 2019 Jul 18. PMID 31326117